CLINICAL TRIAL: NCT03849560
Title: A Multicenter, Double-Blind, Randomized, Parallel Group Study of Safety, Reactogenicity, Immunogenicity, and Efficacy of Quadrivalent Influenza Vaccine Grippol Quadri and Trivalent Influenza Vaccine Grippol Plus in Volunteers.
Brief Title: Safety, Reactogenicity, Immunogenicity, Efficacy of Influenza Vaccines Grippol® Quadri and Grippol® Plus in Volunteers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GriQv-III-16
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grippol® Quadri (Experimental): Grippol® Quadri, a quadrivalent inactivated subunit influenza vaccine. Dosage form: suspension for intramuscular and subcutaneous injection. Dosage: 0.5 ml (1 dose)
  Active ingredients:
  * type A (H1N1) influenza virus antigen 5 µg;
  * type A (H3N2) influenza virus antigen 5 µg;
  * type B (Yamagata lineage) influenza virus antigen 5 µg;
  * type B (Victoria lineage) influenza virus antigen 5 µg;
  * immunoadjuvant Polyoxidonium® (azoximer bromide) 500 µg.
  Interventions: Biological: Grippol® Quadri
- Grippol® Plus, trivalent (Yamagata lineage) (Active Comparator): Grippol® Plus, trivalent inactivated polymer-subunit influenza vaccine containing Yamagata lineage type B influenza virus antigen.
  Dosage form: suspension for intramuscular and subcutaneous injection. Dosage: 0.5 ml (1 dose)
  Active ingredients:
  * type A (H1N1) influenza virus antigen 5 µg;
  * type A (H3N2) influenza virus antigen 5 µg;
  * type B (Yamagata lineage) influenza virus antigen 5 µg;
  * immunoadjuvant Polyoxidonium® (azoximer bromide) 500 µg.
  Interventions: Biological: Grippol® Plus, trivalent (Yamagata lineage)
- Grippol® Plus, trivalent (Victoria lineage) (Active Comparator): Grippol® Plus, trivalent inactivated polymer-subunit influenza vaccine containing Victoria lineage type B influenza virus antigen.
  Dosage form: suspension for intramuscular and subcutaneous injection. Dosage: 0.5 ml (1 dose)
  Active ingredients:
  * type A (H1N1) influenza virus antigen 5 µg;
  * type A (H3N2) influenza virus antigen 5 µg;
  * type B (Victoria lineage) influenza virus antigen 5 µg;
  * immunoadjuvant Polyoxidonium® (azoximer bromide) 500 µg.
  Interventions: Biological: Grippol® Plus, trivalent (Victoria lineage)

INTERVENTIONS:
Biological: Grippol® Quadri — Single intramuscular injection of 0.5 ml (1 dose) of vaccine Grippol® Quadri into the upper third of the outer surface of the shoulder (the deltoid muscle).
  Arms: Grippol® Quadri
Biological: Grippol® Plus, trivalent (Yamagata lineage) — Single intramuscular injection of 0.5 ml (1 dose) of vaccine Grippol® Plus, trivalent (Yamagata lineage) into the upper third of the outer surface of the shoulder (the deltoid muscle).
  Arms: Grippol® Plus, trivalent (Yamagata lineage)
Biological: Grippol® Plus, trivalent (Victoria lineage) — Single intramuscular injection of 0.5 ml (1 dose) of vaccine Grippol® Plus, trivalent (Victoria lineage) into the upper third of the outer surface of the shoulder (the deltoid muscle).
  Arms: Grippol® Plus, trivalent (Victoria lineage)

SUMMARY:
The aim of the study to assess the safety, reactogenicity, immunogenicity, and efficacy of quadrivalent inactivated subunit influenza vaccine Grippol® Quadri (NPO Petrovax Pharm, LLC, Russia) versus trivalent inactivated polymer-subunit vaccine Grippol® Plus (NPO Petrovax Pharm, LLC, Russia) in subjects from 18 to 60 years old.

DETAILED DESCRIPTION:
The first Russian quadrivalent influenza vaccine was developed to improve the effectiveness of vaccination and the cost-effectiveness of preventive immunization.

Task of the study:

1. Study and comparative assessment of the immunogenicity of the influenza quadrivalent inactivated subunit Grippol® Quadri vaccine in comparison with the trivalent inactivated polymer-subunit influenza vaccine Grippol® plus in volunteers aged 18-60 years.
2. Evaluation of the safety and reactogenicity of the influenza quadrivalent inactivated subunit Grippol® Quadri vaccine in comparison with the trivalent inactivated polymer-subunit influenza vaccine Grippol® plus in volunteers aged 18-60 years.
3. Study and comparative evaluation of the efficacy of the influenza quadrivalent inactivated subunit Grippol® Quadri vaccine in comparison with the trivalent inactivated polymer-subunit influenza vaccine Grippol® plus in volunteers aged 18-60 years.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated volunteer's informed consent for participation in the study.
2. Men and women from 18 to 60 years old.
3. Healthy volunteers without signs of acute or chronic disorders, without history of chronic respiratory, cardiovascular, nervous system disorders, hepatic or renal disorders.
4. Previously not immunized, or previous influenza immunization occurring ≥ 12 months before this study.
5. Subjects without history of influenza within ≥ 12 months before this study.
6. Consent of volunteers (men and women) to use adequate methods of contraception (cervical caps with spermicide, diaphragms with spermicide, condoms with spermicide, intrauterine devices, oral contraceptives) or full abstinence for the whole period of the study.

Specific:

1. Contraindications listed in the protocol and prescribing information for inactivated influenza vaccines:

   * acute infections and non-communicable disorders, including the period of reconvalescence of at least one month from the time of clinical and laboratory evidence of recovery;
   * hepatitis or meningococcal infection occurred less than 6 months after recovery;
   * exacerbations of chronic disorder or decompensated disorders that may impact the study (organic central nervous system disorders, decompensated cardiovascular disorder, acute renal or hepatic failure);
   * malignant neoplasms (including hematological disorders);
   * primary immunodeficiency (laboratory-confirmed);
   * HIV infection or HIV-associated disorders;
   * systemic disorders of connective tissue;
   * haemophilia (and other blood coagulation disorders);
   * severe neurological disorders;
   * Guillain-Barré syndrome (post infection demyelinating polyradiculoneuropathy of autoimmune nature with peripheral limb muscle palsy related to inflammation and destruction of myelin sheath of peripheral nerves; may acquire an ascending nature, involving muscles of face, pharynx, larynx);
   * history of severe vaccine-associated reactions (body temperature exceeding 38.5 °С) or local reactions (hyperemia and/or oedema at the site of injection of over 5 cm in diameter);
   * history of severe allergic disorders (angioedema, polymorphic exudative erythema, serum disease, etc.);
   * hypersensitivity to chicken protein or vaccine components;
   * blood and components transfusion within the last 6 months.
2. Indications for immunomodulating therapy.
3. Body temperature over 37.0 °С at screening or before injection.
4. Potential evidence of a chronic infection (periodic episodes of fever within the last 6 months), or antiviral (and/or antibacterial) treatment indicated.
5. History of disorders or conditions, which, according to investigator's judgment may impact the thermal regulation (chronic infections, neuroendocrine disorders [thyrotoxicosis, pheochromocytoma, etc.], climacteric syndrome, malignant hyperthermia, diseases of the central nervous system, malignant neoplasm, connective tissue disorders, systemic vasculitis, and information on excessive physical stress or work-rest regimen deviations [within the last 2 months: night shifts, significant change of time zones, overheating]).
6. Use of antipyretics (including non-steroidal anti-inflammatory drugs and anilides) within 24 hours before randomization.
7. Surgical interventions within less than 90 days before the screening visit.
8. Systolic blood pressure of over 130 mm Hg or less than 100 mm Hg and/or diastolic blood pressure of over 90 mm Hg or less than 60 mm Hg.
9. Any other disorder, which, in the opinion of the investigator, may prevent inclusion of the volunteer due to safety reasons or may impact the study results.

   General:
10. Pregnant and nursing women.
11. Lack of ability to visit daytime inpatient facility according to the study schedule, unavailability for adequate follow-up of the volunteer.
12. Body mass index of less than 18.5 or over 30.0 kg/m2 based on the weight-height Quetelet's index.
13. Participation in another clinical study of medicinal drugs within 3 months before the start of this study.
14. Mental, physical, or other reasons which prevent adequate assessment of own behavior and prevent from meeting the study protocol conditions.
15. History of narcotic and/or drug abuse, and/or inhalant addiction, current signs of alcoholic intoxication.
16. Intake of at least 5 alcohol units per week or history of alcohol, drug, or medicinal product abuse. One alcohol unit corresponds to 360 ml of beer, 120 ml of wine, or 30 ml of a strong alcoholic beverage.
17. Suspected lack of compliance with treatment or inability to undergo treatment and observe the limitations according to the study protocol.
18. Volunteers acknowledged by the court to be disabled or under guardianship.
19. Any other conditions that make the volunteer ineligible for the study according to a justified opinion of the study doctor or Sponsor.

Exclusion Criteria:

* Informed consent recall.
* Occurrence of a severe adverse events (AE) or serious adverse events.
* The volunteer is found to meet any of the non-inclusion criteria related to the safety of the volunteer participation in the study.
* If a female-volunteer becomes pregnant.
* The volunteer takes medicines not allowed in this study.
* The volunteer is lost to follow-up.
* In a situation, which, to the investigator's judgment, may adversely impact the volunteer if he/she continues participating in the study.
* For administrative reasons (study termination by the Sponsor or regulatory authorities) or in case of major protocol violations which may significantly impact the study results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 612 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Chirun, PhD, Study Director — NPO Petrovax; Dmitri Lioznov, PhD, Principal Investigator — Federal State Budgetary Educational Institution of Higher Education "First St. Petersburg State Medical University named after academician I.P. Pavlova "of the Ministry of Health of the Russian Federation.
Locations (3):
- Russia (3):
  - Federal State Budgetary Educational Institution of Higher Education "First St. Petersburg State Medical University named after academician I.P. Pavlova "of the Ministry of Health of the Russian Federation., Saint Petersburg, Leningradskaya Oblast'
  - Federal State Budgetary Institution "Children's Scientific and Clinical Center for Infectious Diseases of the Federal Medical and Biological Agency", Saint Petersburg, Leningradskaya Oblast'
  - Smorodintsev Research Institute of Influenza, Saint Petersburg, Leningradskaya Oblast'

RESULTS

PARTICIPANT FLOW:
Groups:
- Grippol® Quadri: Grippol® Quadri, a quadrivalent inactivated subunit influenza vaccine. Dosage form: suspension for intramuscular and subcutaneous injection. Dosage: 0.5 ml (1 dose)
  Active ingredients:
  * type A (H1N1) influenza virus antigen 5 µg;
  * type A (H3N2) influenza virus antigen 5 µg;
  * type B (Yamagata lineage) influenza virus antigen 5 µg;
  * type B (Victoria lineage) influenza virus antigen 5 µg;
  * immunoadjuvant Polyoxidonium® (azoximer bromide) 500 µg.
  Grippol® Quadri: Single intramuscular injection of 0.5 ml (1 dose) of vaccine Grippol® Quadri into the upper third of the outer surface of the shoulder (the deltoid muscle).
- Grippol® Plus, Trivalent (Yamagata Lineage): Grippol® Plus, trivalent inactivated polymer-subunit influenza vaccine containing Yamagata lineage type B influenza virus antigen.
  Dosage form: suspension for intramuscular and subcutaneous injection. Dosage: 0.5 ml (1 dose)
  Active ingredients:
  * type A (H1N1) influenza virus antigen 5 µg;
  * type A (H3N2) influenza virus antigen 5 µg;
  * type B (Yamagata lineage) influenza virus antigen 5 µg;
  * immunoadjuvant Polyoxidonium® (azoximer bromide) 500 µg.
  Grippol® Plus, trivalent (Yamagata lineage): Single intramuscular injection of 0.5 ml (1 dose) of vaccine Grippol® Plus, trivalent (Yamagata lineage) into the upper third of the outer surface of the shoulder (the deltoid muscle).
- Grippol® Plus, Trivalent (Victoria Lineage): Grippol® Plus, trivalent inactivated polymer-subunit influenza vaccine containing Victoria lineage type B influenza virus antigen.
  Dosage form: suspension for intramuscular and subcutaneous injection. Dosage: 0.5 ml (1 dose)
  Active ingredients:
  * type A (H1N1) influenza virus antigen 5 µg;
  * type A (H3N2) influenza virus antigen 5 µg;
  * type B (Victoria lineage) influenza virus antigen 5 µg;
  * immunoadjuvant Polyoxidonium® (azoximer bromide) 500 µg.
  Grippol® Plus, trivalent (Victoria lineage): Single intramuscular injection of 0.5 ml (1 dose) of vaccine Grippol® Plus, trivalent (Victoria lineage) into the upper third of the outer surface of the shoulder (the deltoid muscle).
Period: Overall Study
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
Started | 205 | 205 | 202
Completed | 204 | 205 | 202
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 612 patients were randomized, 1 patient dropped out during the trial (due to withdrawal of informed consent), data of these patients were used for safety analysis. 611 patients completed the study, data from 607 participants were accepted for the final analysis of immunological efficacy (4 patients were excluded from the analysis due to lack of baseline values for analysis of immunological efficacy), data from 609 participants were used for analysis of secondary outcome measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage) | Total
Number analyzed (Participants) | 205 | 205 | 202 | 612
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.37 (10.15) | 28.97 (10.48) | 29.29 (10.55) | 28.87 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 110 | 111 | 335
  Male | 91 | 95 | 91 | 277
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 205 | 205 | 202 | 612
Height [Mean (Standard Deviation); unit: centimeters] | 171.9 (9.18) | 172.0 (9.28) | 172.3 (9.45) | 172.1 (9.29)
Weight [Mean (Standard Deviation); unit: kilograms] | 68.3 (12.23) | 68.7 (12.41) | 68.7 (11.97) | 68.5 (12.19)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 22.97 (2.86) | 23.09 (2.90) | 23.04 (3.08) | 23.03 (2.94)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Achieving Seroconversion Increased More Than 4-fold Versus Baseline for Antigens: Influenza Virus Type А - H1N1, Influenza Virus Type А - H3N2, Influenza Virus Type В - Yamagata and Victoria Lineage
Description: Percent of subjects achieving seroconversion (the number of volunteers with antibody titer [of at least 1:40] increased more than 4-fold versus baseline [assessed by HAIR]) for antigens: influenza virus type А - H1N1, influenza virus type А - H3N2, influenza virus type В - Yamagata and Victoria lineage, based on assessment at Visit 7.
Time Frame: Day 21 after immunization (Visit 7)
Population: 612 patients were randomized, 1 people dropped out during the trial (due to withdrawal of informed consent). 611 patients completed the study, data from 607 participants were accepted for the final analysis of efficacy (4 patients were excluded from the analysis due to the lack of baseline values for analysis of immunological efficacy).
Measure: Count of Participants; unit: Participants
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
Number analyzed (Participants) | 202 | 203 | 202
Participants
  H1N1 | 133 | 127 | 126
  H3N2 | 140 | 123 | 127
  Victoria (VICT) | 137 | 38 | 127
  Yamagata (YAMA) | 132 | 121 | 59
Statistical Analysis 1: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Yamagata Lineage) vs Grippol® Plus, Trivalent (Victoria Lineage); Test type: Non-Inferiority — Odds ratio was calculated to compare seroconversion for antigen H1N1 in group Grippol® Quadri and groups Grippol® Plus, trivalent (Yamagata lineage)+Grippol® Plus, trivalent (Victoria lineage); Odds Ratio, log = 1.22, 95% CI 2-sided [0.82 to 1.82]
Statistical Analysis 2: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Yamagata Lineage) vs Grippol® Plus, Trivalent (Victoria Lineage); Test type: Non-Inferiority — Odds ratio was calculated to compare seroconversion for antigen H3N2 in group Grippol® Quadri and groups Grippol® Plus, trivalent (Yamagata lineage)+Grippol® Plus, trivalent (Victoria lineage); Odds Ratio, log = 1.54, 95% CI 2-sided [1.08 to 2.30]
Statistical Analysis 3: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Yamagata Lineage); Test type: Non-Inferiority — Odds ratio was calculated to compare seroconversion for YAMA antigen in group Grippol® Quadri and group Grippol® Plus, trivalent (Yamagata lineage); Odds Ratio, log = 1.39, 95% CI 2-sided [0.90 to 2.15]
Statistical Analysis 4: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Victoria Lineage); Test type: Non-Inferiority — Odds ratio was calculated to compare seroconversion for VICT antigen in group Grippol® Quadri and group Grippol® Plus, trivalent (Victoria lineage); Odds Ratio, log = 1.05, 95% CI 2-sided [0.68 to 1.63]

2. Secondary Outcome: Geometric Mean of Serum Antibodies
Description: To antigens: influenza virus type А - H1N1, influenza virus type А - H3N2, influenza virus type В - Yamagata and Victoria lineage.
  Based on assessment at Visit 7.
Time Frame: Day 21 after immunization (Visit 7)
Population: 612 patients were randomized, 1 patient dropped out during the trial, data of these patients were used for safety analysis. 611 patients completed the study (FAS), data from 607 participants were accepted for the final analysis of immunological efficacy - primary outcome measure (4 patients were excluded from the analysis due to lack of baseline values for analysis of immunological efficacy), data from 609 participants were used for analysis of secondary outcome measures.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
Number analyzed (Participants) | 203 | 204 | 202
Titers
  H1N1 | 102.30 [89.54 to 116.95] | 87.39 [76.75 to 99.77] | 94.32 [82.60 to 107.65]
  H3N2 | 70.99 [60.95 to 82.60] | 56.95 [48.98 to 66.22] | 62.06 [53.33 to 72.28]
  VICT | 41.39 [35.97 to 47.53] | 17.05 [14.83 to 19.59] | 47.65 [41.40 to 54.83]
  YAMA | 65.63 [57.15 to 75.51] | 52.85 [46.03 to 60.67] | 34.87 [30.34 to 40.09]
Statistical Analysis 1: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Yamagata Lineage) vs Grippol® Plus, Trivalent (Victoria Lineage); Non-inferiority of Grippol® Quadri over Grippol® Plus, trivalent (Yamagata lineage) and Grippol® Plus, trivalent (Victoria lineage) for the strain A/H1N1; Test type: Non-Inferiority — The Grippol® Quadri vaccine considered non-inferior to Grippol® Plus, trivalent (Yamagata lineage) and Grippol® Plus, trivalent (Victoria lineage) vaccines for the strain A/H1N1 if the upper limit of the two-sided 95% Confidence Interval (CI) of the ratio of means of geometric antibody titers for H1N1 was ≤1.5; Mean Difference (Final Values) = 0.8933, 95% CI 2-sided [0.7762 to 1.030]
Statistical Analysis 2: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Yamagata Lineage) vs Grippol® Plus, Trivalent (Victoria Lineage); Non-inferiority of Grippol® Quadri over Grippol® Plus, trivalent (Yamagata lineage) and Grippol® Plus, trivalent (Victoria lineage) for the strain A/H3N2; Test type: Non-Inferiority — The Grippol® Quadri vaccine considered non-inferior to Grippol® Plus, trivalent (Yamagata lineage) and Grippol® Plus, trivalent (Victoria lineage) vaccines for the strain A/H3N2 if the upper limit of the two-sided 95% CI of the ratio of means of geometric antibody titers for H3N2 was ≤1.5; Median Difference (Final Values) = 0.8913, 95% CI 2-sided [0.7516 to 1.0593]
Statistical Analysis 3: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Yamagata Lineage); Non-inferiority of Grippol® Quadri over Grippol® Plus, trivalent (Yamagata lineage) for the strain B/Yamagata; Test type: Non-Inferiority — The Grippol® Quadri vaccine considered non-inferior to Grippol® Plus, trivalent (Yamagata lineage) vaccine for the strain B/Yamagata if the upper limit of the two-sided 95% CI of the ratio of means of geometric antibody titers for Yamagata antigen was ≤1; Mean Difference (Final Values) = 0.8185, 95% CI 2-sided [0.6918 to 0.9683]
Statistical Analysis 4: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Victoria Lineage); Non-inferiority of Grippol® Quadri over Grippol® Plus, trivalent (Victoria lineage) for the strain B/Victoria; Test type: Non-Inferiority — The Grippol® Quadri vaccine considered non-inferior to Grippol® Plus, trivalent (Victoria lineage) vaccine for the strain B/Victoria if the upper limit of the two-sided 95% CI of the ratio of means of geometric antibody titers for Victoria antigen was ≤1; p = 0.05, ANCOVA; Mean Difference (Final Values) = 1.0328, 95% CI 2-sided [0.8570 to 1.2445]

3. Secondary Outcome: Seroprotection: Percent of Subjects Achieving Protective Antibody Titer (1:40 and More) to Antigens H1N1, H3N2, Yamagata and Victoria Lineage, Based on Assessment at Day 21 After Immunization (Visit 7).
Description: Antibody titer is determined using the hemagglutination inhibition reaction (HAIR), the method recommended by the World Health Organization (WHO) for influenza vaccine efficacy evaluation. As an additional method for 150 volunteers (50 volunteers in each group), a microneutralization assay is planned (the data will be used to evaluate seroprotection). Seroprotection: share of subjects achieving protective antibody titer (1:40 and more, assessed by HAIR and microneutralization test) to antigens H1N1, H3N2, Yamagata and Victoria lineages.
Time Frame: Day 21 after immunization (Visit 7)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
Number analyzed (Participants) | 203 | 204 | 202
Participants
  H1N1 before vaccination (Baseline) | 84 | 86 | 81
  H1N1 day 21 after vaccination | 185 | 184 | 189
  H3N2 before vaccination (Baseline) | 48 | 35 | 48
  H3N2 day 21 after vaccination | 168 | 152 | 168
  Yamagata before vaccination (Baseline) | 55 | 52 | 62
  Yamagata day 21 after vaccination | 173 | 166 | 115
  Victoria before vaccination (Baseline) | 11 | 27 | 27
  Victoria day 21 after vaccination | 154 | 61 | 156
Statistical Analysis 1: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Yamagata Lineage) vs Grippol® Plus, Trivalent (Victoria Lineage); Test type: Non-Inferiority — Seroprotection for strain A/H1N1 in Grippol® Quadri group in comparison to Grippol® Plus, trivalent (Yamagata lineage)+Grippol® Plus, trivalent (Victoria lineage) groups; p = 0.758, Fisher Exact
Statistical Analysis 2: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Yamagata Lineage); Test type: Non-Inferiority — Seroprotection for strain A/H3N2 in Grippol® Quadri group in comparison to Grippol® Plus, trivalent (Yamagata lineage)+Grippol® Plus, trivalent (Victoria lineage) groups; p = 0.282, Fisher Exact
Statistical Analysis 3: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Yamagata Lineage); Test type: Non-Inferiority — Seroprotection for strain B/Yamagata in Grippol® Quadri group in comparison to Grippol® Plus, trivalent (Yamagata lineage) group; p = 0.352, Fisher Exact
Statistical Analysis 4: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Victoria Lineage); Test type: Non-Inferiority — Seroprotection for strain B/Victoria in Grippol® Quadri group in comparison to Grippol® Plus, trivalent (Victoria lineage) group; p = 0.815, Fisher Exact

4. Secondary Outcome: Incidence of Influenza and Acute Respiratory Infection (ARI)
Description: Incidence of influenza and acute respiratory infection (ARI) based on assessment at Visit 11.
Time Frame: Day 180±5 after immunization (Visit 11)
Population: 612 patients were randomized, 1 patient dropped out during the trial (due to withdrawal of informed consent).There were data for this parametr only from 610 patients (1 patient dropped out during the trial, data for another patient is absent for unknown reason).
Measure: Count of Participants; unit: Participants
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
Number analyzed (Participants) | 204 | 204 | 202
Participants | 66 | 59 | 61
Statistical Analysis 1: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Yamagata Lineage); Test type: Other; p = 0.452, Log Rank
Statistical Analysis 2: Comparison: Grippol® Quadri vs Grippol® Plus, Trivalent (Victoria Lineage); Test type: Other; p = 0.639, Log Rank

5. Secondary Outcome: The Average Value of the Total Duration of the Disease in Patients With Acute Respiratory Viral Infections or Influenza in Days .
Description: A case of influenza and ARI is considered as a case of flu-like symptoms (according to: European center for Disease Prevention and Control (ECDC) TECHNICAL DOCUMENT Protocol for case-control studies to measure pandemic and seasonal influenza vaccine effectiveness in the European Union and European Economic Area Member States/ ECDC, 2009): if a subject seeks physician's advice regarding unexpected occurrence of at least one of 4 systemic symptoms: 1) chills or fever, 2) distress, 3) headache, 4) myalgia and at least one of 3 respiratory symptoms: 1) cough, 2) sore throat, 3) respiratory distress.
  Study doctor will perform evaluation of influenza or ARI duration and severity, making phone calls to subject. A case with at least 1 of the complications listed below will be considered severe: the necessity of hospitalization; influenza-associated pneumonia; influenza-associated cardiovascular disorder; death.
Time Frame: Day 180±5 after immunization (Visit 11)
Population: Overall Number of Participants Analyzed here represents the number of participants with incidence of Influenza and ARI
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
Number analyzed (Participants) | 66 | 59 | 61
days | 7.00 (4.743) | 8.05 (5.350) | 9.61 (7.086)

6. Secondary Outcome: Fold Change in Geometric Mean Titer of Serum Antibodies
Description: Fold Change in Geometric Mean Titer of Serum Antibodies (antigens H1N1,H3N2, Yamagata and Victoria lineages) based on assessment data at visit 7.
Time Frame: 21 days following vaccination (visit 7).
Population: 612 patients were randomized, 1 patient dropped out during the trial, data of these patients were used for safety analysis. 611 patients completed the study, data from 607 participants were accepted for the final analysis of immunological efficacy - primary outcome measure (4 patients were excluded from the analysis due to lack of baseline values for analysis of immunological efficacy), data from 609 participants were used for analysis of secondary outcome measures.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of geometric means
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
Number analyzed (Participants) | 203 | 204 | 202
Ratio of geometric means
  H1N1 | 4.86 [4.22 to 5.60] | 4.21 [3.59 to 4.94] | 4.60 [3.97 to 5.34]
  H3N2 | 5.32 [4.53 to 6.24] | 5.22 [4.45 to 6.12] | 5.17 [4.38 to 6.12]
  VICT | 4.77 [4.14 to 5.49] | NA [NA to NA] — Grippol® Plus, trivalent (Yamagata lineage) didn't contain Victoria lineage | 4.72 [4.00 to 5.56]
  YAMA | 5.47 [4.78 to 6.25] | 4.04 [3.48 to 4.96] | NA [NA to NA] — Grippol® Plus, trivalent (Victoria lineage) didn't contain Yamagata lineage
Statistical Analysis 1: Comparison: Grippol® Quadri; Coefficient of increase of mean geometric antibody titer for H1N1 in Grippol® Quadri group; Test type: Other — The lower limit of the two-sided 95% CI (log 10) on coefficient of increase of mean geometric antibody titer for H1N1 should be ˃ 2.5; Coefficient of increase of mean geometri = 4.86, 95% CI 2-sided [4.22 to 5.60]
Statistical Analysis 2: Comparison: Grippol® Quadri; Coefficient of increase of mean geometric antibody titer for H3N2 in Grippol® Quadri group; Test type: Other — The lower limit of the two-sided 95% CI (log 10) on coefficient of increase of mean geometric antibody titer for H3N2 should be ˃ 2.5; Coefficient of increase of GMT = 5.32, 95% CI 2-sided [4.53 to 6.24]
Statistical Analysis 3: Comparison: Grippol® Quadri; Coefficient of increase of mean geometric antibody titer for Yamagata in Grippol® Quadri group; Test type: Other — The lower limit of the two-sided 95% CI (log 10) on coefficient of increase of mean geometric antibody titer for Yamagata should be ˃ 2.5; Coefficient of increase of GMT = 5.47, 95% CI 2-sided [4.78 to 6.25]
Statistical Analysis 4: Comparison: Grippol® Quadri; Coefficient of increase of mean geometric antibody titer for Victoria in Grippol® Quadri group; Test type: Other — The lower limit of the two-sided 95% CI (log 10) on coefficient of increase of mean geometric antibody titer for Victoria should be ˃ 2.5; Coefficient of increase of GMT = 4.77, 95% CI 2-sided [4.14 to 5.49]
Statistical Analysis 5: Comparison: Grippol® Plus, Trivalent (Yamagata Lineage); Coefficient of increase of mean geometric antibody titer for H1N1 in Grippol® Plus, trivalent (Yamagata lineage) group; Test type: Other — [test comment as in outcome 6, analysis 1]; Coefficient of increase of GMT = 4.21, 95% CI 2-sided [3.59 to 4.94]
Statistical Analysis 6: Comparison: Grippol® Plus, Trivalent (Yamagata Lineage); Coefficient of increase of mean geometric antibody titer for H3N2 in Grippol® Plus, trivalent (Yamagata lineage) group; Test type: Other — [test comment as in outcome 6, analysis 2]; Coefficient of increase of GMT = 5.22, 95% CI 2-sided [4.45 to 6.12]
Statistical Analysis 7: Comparison: Grippol® Plus, Trivalent (Yamagata Lineage); Coefficient of increase of mean geometric antibody titer for Yamagata in Grippol® Plus, trivalent (Yamagata lineage) group; Test type: Other — [test comment as in outcome 6, analysis 3]; Coefficient of increase of GMT = 4.04, 95% CI 2-sided [3.48 to 4.69]
Statistical Analysis 8: Comparison: Grippol® Plus, Trivalent (Victoria Lineage); Coefficient of increase of mean geometric antibody titer for H1N1 in Grippol® Plus, trivalent (Victoria lineage) group; Test type: Other — [test comment as in outcome 6, analysis 1]; Coefficient of increase of GMT = 4.60, 95% CI 2-sided [3.97 to 5.34]
Statistical Analysis 9: Comparison: Grippol® Plus, Trivalent (Victoria Lineage); Coefficient of increase of mean geometric antibody titer for H3N2 in Grippol® Plus, trivalent (Victoria lineage) group; Test type: Other — [test comment as in outcome 6, analysis 2]; Coefficient of increase of GMT = 5.17, 95% CI 2-sided [4.38 to 6.12]
Statistical Analysis 10: Comparison: Grippol® Plus, Trivalent (Victoria Lineage); Coefficient of increase of mean geometric antibody titer for Victoria in Grippol® Plus, trivalent (Victoria lineage) group; Test type: Other — [test comment as in outcome 6, analysis 4]; Coefficient of increase of GMT = 4.72, 95% CI 2-sided [4.00 to 5.56]

7. Secondary Outcome: Severity of Reported Cases of Influenza and ARI.
Description: A case of influenza and ARI is considered as a case of flu-like symptoms (according to: ECDC TECHNICAL DOCUMENT Protocol for case-control studies to measure pandemic and seasonal influenza vaccine effectiveness in the European Union and European Economic Area Member States/ European center for Disease Prevention and Control, 2009): if a subject seeks physician's advice regarding unexpected occurrence of at least one of 4 systemic symptoms: 1) chills or fever, 2) distress, 3) headache, 4) myalgia and at least one of 3 respiratory symptoms: 1) cough, 2) sore throat, 3) respiratory distress.
  Study doctor will perform evaluation of influenza or ARI duration and severity, making phone calls to subject. A case with at least 1 of the complications listed below will be considered severe: the necessity of hospitalization; influenza-associated pneumonia; influenza-associated cardiovascular disorder; death.
Time Frame: Day 180±5 after immunization (Visit 11)
Population: Overall Number of Participants Analyzed here represents the number of participants with incidence of Influenza and ARI
Measure: Count of Participants; unit: Participants
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
Number analyzed (Participants) | 66 | 59 | 61
Participants
  mild | 60 | 54 | 51
  moderate | 6 | 5 | 10

8. Secondary Outcome: Average Time (Months) to the First Reported Episode of Influenza and ARI
Description: Average time (months) to the first reported episode of influenza and ARI based on assessment at Visit 11.
Time Frame: Day 180±5 after immunization (Visit 11)
Population: 612 patients were randomized, 1 patient dropped out during the trial (due to withdrawal of informed consent).There were data for this parameter only from 610 patients (1 patient dropped out during the trial, data for another patient is absent for unknown reason).
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
Number analyzed (Participants) | 204 | 204 | 202
months | 4.626 [4.319 to 4.934] | 5.111 [4.836 to 5.385] | 4.819 [4.529 to 5.110]

9. Secondary Outcome: Seroprotection: Percent of Subjects Achieving Protective Antibody Titer (1:40 and More) to Antigens H1N1, H3N2, Yamagata and Victoria Lineage, Based on Assessment at Day 21 After Immunization (Additional Method of Analysis: a Microneutralization Assay)
Description: As an additional method for 149 volunteers, a microneutralization assay is planned (the data will be used to evaluate seroprotection). Seroprotection: share of subjects achieving protective antibody titer (1:40 and more, assessed by HAIR and microneutralization test) to antigens H1N1, H3N2, Yamagata and Victoria lineages.
Time Frame: Day 21 after immunization (Visit 7)
Population: Additional method of analysis only for 149 volunteers
Measure: Count of Participants; unit: Participants
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
Number analyzed (Participants) | 51 | 51 | 47
Participants
  H1N1 | 31 | 23 | 27
  H3N2 | 31 | 26 | 34
  Yamagata | 29 | 20 | 13
  Victoria | 26 | 10 | 26

10. Secondary Outcome: Number of Participants With Symptoms of Influenza and ARI in Vaccination Groups
Description: The presence of ARI symptoms in participants in each group is assessed throughout the study. The presence of a symptom at least once is taken into account in the analysis if the participant has several filling out of the questionnaire.
Time Frame: Day 180±5 (Visit 11)
Population: Overall Number of Participants Analyzed here represents the number of participants with incidence of Influenza and ARI;
Measure: Count of Participants; unit: Participants
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
Number analyzed (Participants) | 66 | 59 | 61
Participants
  Sore throat | 41 | 41 | 39
  Headache | 27 | 24 | 28
  Respiratory difficulty | 38 | 40 | 38
  Cough | 30 | 18 | 28
  Myalgia | 5 | 1 | 5
  Feeling of being unwell | 61 | 56 | 56
  Chills or fever | 19 | 22 | 21

ADVERSE EVENTS:
Time Frame: 180±5 Days
Description: No serious adverse events (SAE) or AEs leading to withdrawal from the study were reported after phase 1 study. There were no cases of SAE or death during the current phase 2-3 study.
Arm/Group | Grippol® Quadri | Grippol® Plus, Trivalent (Yamagata Lineage) | Grippol® Plus, Trivalent (Victoria Lineage)
All-Cause Mortality (participants affected / at risk) | 0/205 | 0/205 | 0/202
Serious Adverse Events (participants affected / at risk) | 0/205 | 0/205 | 0/202
Other Adverse Events (participants affected / at risk) | 90/205 | 92/205 | 93/202
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Grippol® Quadri (N=205) | Grippol® Plus, Trivalent (Yamagata Lineage) (N=205) | Grippol® Plus, Trivalent (Victoria Lineage) (N=202)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 3 | 1
Hyperthermia (General disorders) | 0 | 1 | 0
Fever (General disorders) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Furunculosis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Herpes in the nose (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 4 | 4 | 3
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Acute pyelonephritis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 68 | 68 | 74
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 6 | 7 | 4
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Кашель (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT03849560/Prot_SAP_000.pdf